CLINICAL TRIAL: NCT05963243
Title: A Volunteer Study to Collect Imaging Data for the Development of Identifying Probe Pressure as Part of ScanNav Assist Automated Dating Scan
Brief Title: Automated Dating Scan Probe Pressure Data Collection Plan
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2023_WH_02
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy adult (18+ years old) volunteers
  Interventions: Other: Ultrasound Scans

INTERVENTIONS:
Other: Ultrasound Scans — Ultrasound scans collected by experts in ultrasound-guided regional anaesthesia.

SUMMARY:
The goal of this observational study is to collect data in the form of ultrasound recordings from healthy volunteers, to aid the development of an Artificial Intelligence model that can identify ultrasound probe pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

1. Aged <18 years of age;
2. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers from the South Wales region.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Ultrasound scan recordings | 6 months
  Ultrasound scan recordings collected by the volunteer healthy participants of an abdominal self-scan.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Margetts, Dr, Principal Investigator — Intelligent Ultrasound
Locations (1):
- Hodge House, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No